CLINICAL TRIAL: NCT06211296
Title: A Prospective, Multicenter, Non-Randomized, Single-Arm, Open-Label Continued Access Study of the ShortCut™ Device (The ShortCut™ CAS).
Brief Title: The ShortCut™ Continued Access Study Protocol
Acronym: ShortCut-CAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pi-cardia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S01-CLN-023
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Valve-in-valve Procedures; Aortic Stenosis; Coronary; Obstruction
Keywords: TAVI; Pi-Cardia; TAVR; ViV; continued access; Shortcut
MeSH Terms: conditions — Aortic Valve Stenosis; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Shortcut (Experimental): Splitting bioprosthetic aortic valve leaflets
  Interventions: Device: Shortcut

INTERVENTIONS:
Device: Shortcut — Splitting bioprosthetic aortic valve leaflets

SUMMARY:
A Prospective, Multicenter, Non-Randomized, Single-Arm, Open-Label Continued Access Study of the ShortCut™ device (The ShortCut™ CAS).

DETAILED DESCRIPTION:
The continued access study will be used to collect additional safety and effectiveness data of the ShortCut™ device for splitting bioprosthetic aortic valve leaflets, and to demonstrate coronary artery ostia patency following leaflet split, in patients who are at risk for TAVR-induced coronary artery ostium obstruction following a ViV procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is planned to undergo a percutaneous valve-in-valve procedure for an approved ViV indication due to a failed bioprosthetic valve.
2. Patient is at risk for TAVR-induced coronary artery ostium obstruction.
3. Written informed consent to participate in the study obtained from the subject or subject's legal representative, according to local regulations, prior to initiation of any study mandated procedure.

Exclusion Criteria:

1. An excessive aortic valve leaflet Calcium morphology, such as diffuse massive calcification at the targeted leaflet for splitting or anatomy not suitable for the use of the ShortCut™ device, as determined by the CT measurements.
2. Carotid or vertebral artery disease that, in the opinion of the local Heart Team, should be treated; or treatment of carotid stenosis ≤ 1 month prior to index procedure.
3. CVA or TIA ≤ 6 months prior to index procedure.
4. History of a myocardial infarction (MI) ≤ 6 weeks prior to index procedure.
5. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance.
6. LVEF < 30%.
7. Ongoing severe infection or sepsis.
8. Patient has renal insufficiency or is on chronic dialysis.

8. Need for emergency surgery for any reason. 9. Life expectancy is less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Givon, Study Director — Pi-cardia
Locations (4):
- United States (4):
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center /NYPH, New York, New York
  - UPMC Pinnacle, Wormleysburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shortcut
Started | 8
30 Days Follow up | 8
90 Days Follow up | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7
  Unknown | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
STS score [Mean (Standard Deviation); unit: units on a scale] — STS: Society of Thoracic Surgeons (STS) Risk Score - estimates the risk of mortality and major morbidity following cardiac surgery.
  Range: 0% to 100% (represents the predicted probability of death or a major adverse event)
  Typical Range Observed in Clinical Use: Usually <1% to ~20%, depending on procedure and patient risk profile.
  Directionality:
  Higher values = worse outcomes / higher surgical risk
  Lower values = better outcomes / lower surgical risk
  units on a scale | 10.3 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: ShortCut™ Device- and/or ShortCut™ Procedure-related: Mortality, Stroke
Description: Primary safety endpoint, ShortCut™ device- and/or ShortCut™ procedure-related: Mortality, Stroke
Time Frame: discharge or at 7 days post-procedure, whichever occurs first
Measure: Number; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Number of Participants With Leaflet Splitting Success Using the Shortcut Device, Assessed by Echo and/or Angiography
Description: Primary effectiveness endpoint, Leaflet splitting success using the Shortcut Device, assessed by echo and/or angiography
Time Frame: Intra-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 8

3. Secondary Outcome: Rate of All Cause Mortality, Per VARC 3
Description: Secondary safety endpoint, Rate of all cause mortality, per VARC 3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

4. Secondary Outcome: Rate of All-cause Stroke, Per VARC-3
Description: Secondary safety endpoint, Rate of all-cause stroke, per VARC-3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

5. Secondary Outcome: Rate of Coronary Obstruction Per VARC-3
Description: Secondary safety endpoint, Rate of coronary obstruction per VARC-3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

6. Secondary Outcome: Rate of MI With New Evidence of Coronary Artery Obstruction Requiring Intervention Per VARC-3
Description: Secondary safety endpoint, Rate of MI with new evidence of coronary artery obstruction requiring intervention per VARC-3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

7. Secondary Outcome: -Rate of Major Vascular Complications Per VARC-3
Description: Secondary safety endpoint, -Rate of major vascular complications per VARC-3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

8. Secondary Outcome: Rate of Cardiac Temponade Per VARC-3
Description: Secondary safety endpoint, Rate of cardiac temponade per VARC-3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

9. Secondary Outcome: Rate of Acute Kidney Injury Per VARC-3
Description: Secondary safety endpoint, Rate of Acute Kidney Injury per VARC-3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

10. Secondary Outcome: Access-related Type 3-4 Bleeding Per VARC-3
Description: Secondary safety endpoint, Access-related type 3-4 bleeding per VARC-3
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

11. Secondary Outcome: Rate of Freedom From Coronary Artery Intervention Related to the Intervened Leaflet
Description: Secondary effectiveness endpoint, Rate of freedom from coronary artery intervention related to the intervened leaflet
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 8

12. Secondary Outcome: Rate of Freedom From Coronary Artery Ostia Obstruction Related to the Intervened Leaflet
Description: Secondary effectiveness endpoint, Rate of freedom from coronary artery ostia obstruction related to the intervened leaflet
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 8

13. Secondary Outcome: Shortcut Technical Success
Description: Technical success endpoint, Shortcut technical success - Successful access, delivery, and retrieval of the ShortCut™ device.
Time Frame: At exit from procedure room, immediately after the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 7

14. Other Pre Specified Outcome: Rate of All Cause Mortality Per VARC-3
Description: Tertiary Safety Endpoint, Rate of all cause mortality per VARC-3
Time Frame: 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

15. Other Pre Specified Outcome: Rate of Stroke Per VARC-3
Description: Tertiary Safety Endpoint, Rate of stroke per VARC-3
Time Frame: 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

16. Other Pre Specified Outcome: Rate of MI With New Evidence of Coronary Artery Obstruction Requiring Intervention Per VARC-3
Description: Tertiary Safety Endpoint, Rate of MI with new evidence of coronary artery obstruction requiring intervention per VARC-3
Time Frame: 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shortcut
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported from point of index procedure until 90 days post procedure
Arm/Group | Shortcut
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shortcut (N=8)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac standstill (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT06211296/Prot_SAP_002.pdf